CLINICAL TRIAL: NCT02693964
Title: Bone and Vascular Health in Postmenopausal Women With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1854
Record Dates: First submitted 2016-02-18; First posted 2016-02-29 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes; Menopause; Cardiovascular Risk; Bone Density
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Bone Density

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Postmenopausal women with T1D: Postmenopausal between 45-70 years of age and having T1D for at least 10 years
  Interventions: Other: Bone density and carotid ultrasound
- Postmenopausal women without diabetes: Postmenopausal between 45-70 years of age without diabetes
  Interventions: Other: Bone density and carotid ultrasound

INTERVENTIONS:
Other: Bone density and carotid ultrasound — All participants will be asked for relevant medical, personal, family and diabetes history, treatment and complications, and history of falls and fractures and will undergo measurement of bone density, carotid ultrasound and a blood draw.

SUMMARY:
The study is designed to evaluate the differences in bone mineral density (BMD) and Carotid Intima Media Thickness (CIMT) between postmenopausal women with type 1 diabetes (T1D) compared to postmenopausal women without diabetes.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is an autoimmune disease requiring lifelong insulin treatment. Having T1D increases the risk of death, especially in women with T1D.

Heart disease and fractures due to osteoporosis (brittle bones) are the leading causes of death in women with T1D.

Since both diseases share certain common risk factors such as age, menopause, smoking, physical inactivity, and diabetes, this study is designed to find link between bone density and cardiovascular risk.

This study has only one visit. All participants will undergone bone density testing using a dual energy x-ray absorptiometry (DEXA) machine and measurement of carotid intima media thickness (a marker of carotid atherosclerosis) using carotid ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* T1D as defined under CACTI study OR Controls as defined as no current diabetes (HbA1c < 6.5% and fasting blood glucose < 126 mg/dl, no diabetes diagnosis and no use of anti-diabetic medication),
* Diabetes duration of 10 years or greater, and
* Postmenopausal women. Menopause is defined as no menstrual periods for at least 12 consecutive months OR FSH greater than 40 IU/L on at least two occasions.

Exclusion Criteria:

* Chronic diseases, which can affect the BMD measurement such as:

  * Uncontrolled coeliac or thyroid disease,
  * Addison's disease,
  * Malabsorption syndrome,
  * Rheumatologic disorder,
  * Parathyroid disorders,
  * Cancer other than skin cancer, and
  * Chronic kidney disease with eGFR less than 30.
* Medications that can affect BMD results such as:

  * Oral or injectable steroid intake for more than 3 months,
  * Immunosuppressant and osteoanabolic or antiresorptive medications for osteoporosis treatment, and
  * Previous fractures or deformities making it difficult to perform DXA at hip and spine.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with or without type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Difference in bone mineral density between postmenopausal women with type 1 diabetes and controls | at baseline
  Postmenopausal women with T1D will have lower BMD at hip, lumbar spine and distal radius and higher cardiovascular risk as assessed by carotid intima media thickness (CIMT) compared to age and weight matched postmenopausal women without diabetes.
Difference in carotid intima media thickness between postmenopausal women with type 1 diabetes and controls | at baseline
  Postmenopausal women with T1D will have lower BMD at hip, lumbar spine and distal radius and higher cardiovascular risk as assessed by carotid intima media thickness (CIMT) compared to age and weight matched postmenopausal women without diabetes.

SECONDARY OUTCOMES:
Differences in biomarkers (1): e.g. (bone specific alkaline phosphatase, Procollagen I Intact N-Terminal (P1NP), osteocalcin, C-terminal telopeptide (CTX): (Continued in Outcome 4) | at baseline
  Bone markers such as osteocalcin, osteopontin and osteoprotogerin and inflammatory markers such as hs-CRP, IL-2, IL-6 and TNF-α will differ by diabetes status and will be associated with the lower bone density and higher cardiovascular risk in postmenopausal women with T1D.
Differences in biomarkers (2): (Continued from Outcome 3) e.g. IL-2, IL-6 (Interleukin 2 and 6) and Tumor necrosis factor (TNF-alfa) between postmenopausal women with T1D and controls. | at baseline
  Bone markers such as osteocalcin, osteopontin and osteoprotogerin and inflammatory markers such as hs-CRP, IL-2, IL-6 and TNF-α will differ by diabetes status and will be associated with the lower bone density and higher cardiovascular risk in postmenopausal women with T1D.
Correlation between biomarkers with cardiovascular risk measures (carotid intima media thickness) | at baseline
  Postmenopausal women with T1D will have lower BMD at hip, lumbar spine and distal radius and higher cardiovascular risk as assessed by carotid intima media thickness (CIMT) compared to age and weight matched postmenopausal women without diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Viral Shah, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center for Diabetes, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah VN, Shah CS, Snell-Bergeon JK. Type 1 diabetes and risk of fracture: meta-analysis and review of the literature. Diabet Med. 2015 Sep;32(9):1134-42. doi: 10.1111/dme.12734. Epub 2015 Jun 12. PMID 26096918
- [Background] Dhaon P, Shah VN. Type 1 diabetes and osteoporosis: A review of literature. Indian J Endocrinol Metab. 2014 Mar;18(2):159-65. doi: 10.4103/2230-8210.129105. PMID 24741510
- [Background] Shah VN, Joshee P, Sippl R, Pyle L, Vigers T, Carpenter RD, Kohrt W, Snell-Bergeon JK. Type 1 diabetes onset at young age is associated with compromised bone quality. Bone. 2019 Jun;123:260-264. doi: 10.1016/j.bone.2019.03.039. Epub 2019 Mar 29. PMID 30936041